CLINICAL TRIAL: NCT03208361
Title: Efficacy of High Doses of Oral Penicillin V Versus High Doses of Oral Amoxicillin in the Treatment of Non-severe Community-acquired Pneumonia in Adults
Brief Title: Efficacy of High Doses Penicillin V Versus High Doses Amoxicillin in the Treatment of Non-severe Pneumonia.
Acronym: PENIPNEUMO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of financial support to continue with the study recruitment. Independent study financially supported by a national grant with a 4.5 years duration.
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IJG-PEN-2012; 2012-003511-63 (EudraCT Number)
Record Dates: First submitted 2017-06-26; First posted 2017-07-05 (Actual); Last update posted 2017-07-05 (Actual); Status verified 2017-06

CONDITIONS: Community-acquired Pneumonia (CAP)
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Penicillin V; Amoxicillin

STUDY DESIGN:
Intervention Model Description: Arm 1: Penicillin V (phenoxymethylpenicillin) Arm 2: Amoxicillin (control)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Penicillin V (Experimental): Penicillin V, 1600000 IU every 8h during 10 days.
  Interventions: Drug: Penicillin V
- Amoxicillin (Active Comparator): Amoxicillin, 1 g every 8h during 10 days.
  Interventions: Drug: Amoxicillin

INTERVENTIONS:
Drug: Penicillin V
  Arms: Penicillin V
Drug: Amoxicillin
  Arms: Amoxicillin

SUMMARY:
This study aims to evaluate wether high-dose penicillin V is as effective as high-dose amoxicillin for the treatment of non-sever community-acquired pneumonia (CAP).

DETAILED DESCRIPTION:
Phase III parallel-group, randomised, double blind clinical trial, performed in 31 primary healthcare centres in Spain.

The use of narrow-spectrum antibiotics is needed because of the dearth of new antimicrobials and the link observed between the consumption of broad-spectrum antibiotics and the emergence and spread of antibacterial resistance.

Objective: The aim of the present trial was to determine whether high-dose penicillin V was as effective as high-dose amoxicillin for the treatment of uncomplicated CAP in a Mediterranean adult population.

Subjects: Patients between 18-75 years with lower respiratory tract infection and radiologically confirmed diagnosis of pneumonia.

Primary outcome: Clinical resolution at day 14

Visit Schedule: Initiation visit, day 3 phone call, day 14 presential visit, day 30 presential visit.

Quality: The study will be conducted in accordance with the principles of the Declaration of Helsinki, ICH Guidelines for GCP and in full conformity with relevant regulations. The study has been approved by the Ethical Committee of Investigation in Primary Care (Fundació d'Investigació en Atenció Primària) and by the Agencia Española del Medicamento y Productos Sanitarios. The study data was fully monitored by speciallized personnel.

Sample size: The objective of the study is to demonstrate that penicillin V is not inferior to amoxicillin. Considering a success rate of 85% for the group treated with amoxicillin [1,2]. A total of 105 patients will be required in each treatment group (total of 210) to detect a non-inferiority margin of 15% between the two treatments with a minimum power of 80% considering an alpha error of 2.5% for a unilateral hypothesis and maximum possible losses of 15%.

Statistical analyses:The intention-to-treat (ITT) population included all randomized patients receiving at least one dose of study drug and the per-protocol (PP) population included patients who received no systemic antimicrobial agents other than the study drug for at least three days in the case of clinical failure or ≥80% of study medication in the case of cure, with adequate assessment of compliance and absence of major protocol violations.

To evaluate the comparability of the groups the two groups will be analysed with variables expressed as means and standard deviations for the case of quantitative variables and with proportions in the case of qualitative variables. The variable of the principle result, clinical cure, will be expressed as percentages and the comparison of percentages in the two treatment groups will be analysed using the Chi-square test. Logistic regression will be performed for the analysis of the predictive factors of cure or not, with calculation of the odds ratio for each of the variables analysed and multiadjustment for each of the factors of the study with confidence intervals of 95%. Variables with a p<0.20 on bivariant analysis will be included in the analysis. A p value < 0.05 will be considered statistically significant.

The protocol of the study has been published (3)

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years to 75 years (inclusive).
* Signs and symptoms of lower respiratory tract infection.
* Radiological confirmation of the diagnosis of pneumonia or not radiological confirmation but the patient has the following symptoms: high fever (> 38.5 ° C), cough and purulent sputum and auscultation of crackles in a pulmonary focus, the researcher undertakes to confirm after inclusion pneumonia with mandatory radiological study.
* Signature of informed consent.

Exclusion Criteria:

* Impaired consciousness: confused state, delirium, drowsiness, stupor or coma, at the discretion of the investigator
* Respiratory rate> 30 breaths / minute
* Heart rate> 125 beats / minute
* Systolic blood pressure <90 mm ??Hg or diastolic BP <60 mm Hg
* Hypersensitivity to beta-Lactamics
* O2 saturation <92%
* Axillary temperature> 40 ° C
* bronchial Asthma
* Pregnancy or lactation
* Significant comorbidities: renal failure, liver cirrhosis, heart failure, chronic obstructive pulmonary disease, ischemic heart disease diagnosed less than 6 months, stroke diagnosed less than 6 months ago and / or type 1 diabetes mellitus
* Significant alteration in chest radiography: alveolar infiltrates in more than one lobe or bilateral pleural effusion or pulmonary cavitation
* Problems to meet the treatment at home: sociopathy or psychiatric problems, drug and alcohol addiction, or, an unsuitable family environment
* Lack of tolerance to oral therapy: presence of nausea and vomiting, gastrectomy, post-surgery or frank diarrhea
* Immunosuppression: chronic HIV infection, transplant, neutropenic, or, patients receiving immunosuppressive therapy
* active malignancy
* terminal disease
* Hospitalization in the last month
* Taking any systemic antibiotic in the previous three days or a full use of oral antibiotics prior to inclusion in the previous two weeks (use of urinary antiseptics is not a reason for exclusion).
* Difficulty to attend follow-up visits
* Refusal to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-11-05 (Actual); Primary Completion 2016-03-29 (Actual); Study Completion 2016-04-21 (Actual)

PRIMARY OUTCOMES:
Disappearance of fever | 14 days after inclusion
  Disappearance of fever (included in the general definition of Clinical Cure)
Disappearance or improvement of cough | 14 days after inclusion
  Disappearance or improvement of cough (included in the general definition of Clinical Cure)
Improvement of general condition | 14 days after inclusion
  Improvement of general condition (included in the general definition of Clinical Cure)
Disappearance or reduction of auscultation of crackles | 14 days after inclusion
  Disappearance or reduction of auscultation of crackles (included in the general definition of Clinical Cure)
No other antimicrobial treatment necessary | 14 days after inclusion
  No other antimicrobial treatment necessary (included in the general definition of Clinical Cure

SECONDARY OUTCOMES:
Disappearance of fever | 30 days after inclusion
  Disappearance of fever (included in the general definition of Clinical Cure)
disappearance or improvement of cough | 30 days after inclusion
  disappearance or improvement of cough (included in the general definition of clinical cure)
improvement of general condition | 30 days after inclusion
  improvement of general condition (included in the general definition of clinical cure)
disappearance or reduction of auscultation of crackles | 30 days after inclusion
  disappearance or reduction of auscultation of crackles (included in the general definition of clinical cure)
No other antimicrobial treatment necessary | 30 days after inclusion
  No other antimicrobial treatment necessary (included in the general definition of Clinical cure)
Total Clinical Resolution | 14 days after inclusion
  Total resolution of acute signs and symptoms, so no other antimicrobial treatment is needed.
Total Clinical Resolution | 30 days after inclusion
  Total resolution of acute signs and symptoms, so no other antimicrobial treatment is needed.
Radiological resolution | 30 days after inclusion
  Partial or complete resolution of the pulmonar condensation Chest X-Ray
Adverse Events | 1-30 days
  Presence of adverse events during all the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Car Llor Vilà, MD, PhD, Principal Investigator — Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Locations (1):
- IDIAP Jordi Gol, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aubier M, Verster R, Regamey C, Geslin P, Vercken JB. Once-daily sparfloxacin versus high-dosage amoxicillin in the treatment of community-acquired, suspected pneumococcal pneumonia in adults. Sparfloxacin European Study Group. Clin Infect Dis. 1998 Jun;26(6):1312-20. doi: 10.1086/516366. PMID 9636854
- [Background] Petitpretz P, Arvis P, Marel M, Moita J, Urueta J; CAP5 Moxifloxacin Study Group. Oral moxifloxacin vs high-dosage amoxicillin in the treatment of mild-to-moderate, community-acquired, suspected pneumococcal pneumonia in adults. Chest. 2001 Jan;119(1):185-95. doi: 10.1378/chest.119.1.185. PMID 11157603
- [Background] Llor C, Arranz J, Morros R, Garcia-Sangenis A, Pera H, Llobera J, Guillen-Sola M, Carandell E, Ortega J, Hernandez S, Miravitlles M. Efficacy of high doses of oral penicillin versus amoxicillin in the treatment of adults with non-severe pneumonia attended in the community: study protocol for a randomised controlled trial. BMC Fam Pract. 2013 Apr 17;14:50. doi: 10.1186/1471-2296-14-50. PMID 23594463